CLINICAL TRIAL: NCT02541539
Title: Effects of Lactobacillus Casei in the Prevention of Upper Respiratory and Diarrheal Diseases Among Adults
Brief Title: Effects of Lactobacillus Casei on Respiratory and Gastrointestinal Diseases in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Collaborators: Inner Mongolia University of Science and Technology (Other)
Responsible Party: Principal Investigator, Min-Tze LIONG, Associate Professor Dr, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 15020059
Record Dates: First submitted 2015-08-24; First posted 2015-09-04 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus casei Zhang (Active Comparator): Intervention consists of daily administration of 2g probiotic Lactobacillus casei Zhang, administered daily at a fixed dosage of 9 log CFU/sachet/day and continue for 12 months.
  Interventions: Dietary Supplement: Lactobacillus casei Zhang
- Placebo (Placebo Comparator): Intervention consists of daily administration of 2g placebo (no probiotic bacteria), administered daily and continue for 12 months.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lactobacillus casei Zhang — This project aims to study the benefits of probiotics namely Lactobacillus casei Zhang in prevention of upper respiratory and gastrointestinal illnesses, among adults in Malaysia aged from 18-81 years.
  Other Names: LCZ
  Arms: Lactobacillus casei Zhang
Dietary Supplement: Placebo — This project aims to study the benefits of probiotics namely Lactobacillus casei Zhang in prevention of upper respiratory and gastrointestinal illnesses, among adults in Malaysia aged from 18-81 years.
  Arms: Placebo

SUMMARY:
This project aims to study the benefits of probiotics namely Lactobacillus casei Zhang (LCZ) in prevention of upper respiratory and gastrointestinal illnesses, which are found common among adults in Malaysia aged from 18 to 81 years.

DETAILED DESCRIPTION:
Probiotic can be defined as "live microorganisms that grant health effects to the host if consumed in sufficient amounts". Probiotic bacteria, which beneficially affect the host by improving the intestinal microbial balance, may affect the immune response, thus boosting the body system to combat against diseases.

Respiratory tract infections (RTI) can be described as infections on sinuses, throat, airways and lungs. Generally, RTI can be categorized into upper respiratory tract infections (URTI) and lower respiratory tract infections (LRTI). Some of the common URTI are like common cold, sinusitis, pharyngitis, epiglottitis and laryngotracheitis (croup) while examples of LRTI are bronchitis, bronchiolitis and pneumonia. URTI will be the main focus of this research. Despite continuous medical advancement, URTI remains a burden to the vast global communities.In Malaysia, URTI take out a proportion of 16.5% and 21.2% of the diseases diagnosed in public and private health clinics respectively.

Diarrhea is one of the most common symptoms for gastrointestinal diseases. Diarrhea is commonly defined as three or more loose or watery stools in the last 24 hours. Probiotics such as Lactobacillus GG, Bifidobacterium lactis (alone or in combination with Streptococcus thermophiles), and Lactobacillus reuteri, Lactobacillus casei and Lactobacillus acidophilus have been reported to reduce diarrhea-related symptoms in a strain-dependent and dose-dependent manner. The rationale for using probiotics in infectious diarrhoea is that they act against enteric pathogens by competing for available nutrients and binding sites, making the gut contents acid, producing a variety of chemicals, and increasing specific and non-specific immune responses.

Lactobacillus casei Zhang (LCZ) has been identified as a unique probiotic strain that shows favorable probiotic characteristics like high acid and bile tolerance, ability to colonize gastrointestinal tract, in addition to antibacterial, antioxidative and immunomodulatory properties. LCZ was first isolated from koumiss collected in Xilin Guole, Inner Mongolia, China by a group of researchers from Inner Mongolia Agricultural University. Koumiss is a type of fermented horse milk drink which is commonly found in Inner Mongolia, China and has been reported to treat digestive diseases and chronic diseases.

LCZ is already commercially available and currently marketed in China since 2010, in the form of beverages, tablets, powders and capsules. Among the well known products present in the market are Bio-Plus, a type of plant based fermented soymilk beverages, Sci-Plus, and a multiple probiotic tablet. Research and development involving LCZ have won many awards. Among them are 2009 National Science and Technology Progress Award of China (second prize), 2009 Inner Mongolia Natural Science Award (first prize) and the sixth DBN Technology Achievement Award. In addition, up to September 2014, 11 patents were filed and approved while 8 more patents were in the review stage. Besides that, 82 research papers related to LCZ were also published.

Most research on LCZ have been related to improving human's health such as reduce susceptibility to type II diabetes and enhance human's immune system, and also related to food industry usage such as in cheese making industry. More importantly, many of probiotics have been reported to exert health benefits via maintain a healthy gut profile. In a recent clinical study, LCZ was found to significantly altered the composition of intestinal microbiota and the gut microbiota diversity, with a positive correlation with beneficial microorganisms such as Lactobacillus, Bifidobacterium and an unidentified genus from Bacteroidaceae, and a negative correlation with detrimental pathogens such as Clostridium, Serratia, Enterococcus, Shigella and Shewanella, with just a consumption of 28 days.

LCZ has confirmed its safety for consumption, and for this intervention, it will be produced in a HACCP and ISO 22000 certified manufacturing plant (GeneFerm Biotechnology Co., Ltd., Taiwan). LCZ does not contain any porcine or bovine ingredients and has obtained the Halal certification from Taiwan Halal Integrity Development Association (THIDA), Taiwan, which is recognized by Jabatan Kemajuan Islam Malaysia (JAKIM), an organization that oversees the implementation of Halal requirement in Malaysia.

A total number of 150 healthy adults from age 18 -81 years old will be recruited for this study.

ELIGIBILITY:
Inclusion Criteria:

* Male/ female subjects
* 18-81 years old
* Body mass index (BMI) within a healthy range
* Willing to commit throughout the experiment

Exclusion Criteria:

* Type-1 diabetes
* Long term medication due to certain severe illness
* Human immunodeficiency virus/acquired immune deficiency syndrome (HIV/AIDS)
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Vegetarian

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Serum immunoglobulin-A (IgA) level | 12 months
  IgA as an indicator for immunology, in assessing severity of upper respiratory illnesses between number of adult participants taking LCZ vs. placebo
Bristol stool chart scale | 12 months
  Bristol stool scale (from a scale of 1-7; scale of 1 representing hard lump, and 7 representing liquid with no solid pieces) as an indicator for assessing severity of gastrointestinal-related diarrheal illnesses between number of adult participants taking LCZ vs. placebo

SECONDARY OUTCOMES:
Fecal microbiota profiling | 12 months
  Deoxyribonucleic acid (DNA) sequencing of fecal samples to compare DNA sequences of the different microbiota between adult participants taking LCZ vs. placebo

CONTACTS AND LOCATIONS:
Overall Officials: Min tze Liong, PhD, Principal Investigator — USM
Locations (1):
- School of Industrial Technology, Universiti Sains Malaysia, Pulau Pinang, Pulau Pinang, Malaysia

REFERENCES:
- [Result] Zhang J, Wang L, Guo Z, Sun Z, Gesudu Q, Kwok L, Menghebilige, Zhang H. 454 pyrosequencing reveals changes in the faecal microbiota of adults consuming Lactobacillus casei Zhang. FEMS Microbiol Ecol. 2014 Jun;88(3):612-22. doi: 10.1111/1574-6941.12328. PMID 24702028